CLINICAL TRIAL: NCT03169075
Title: Study Evaluating the Feasibility and Efficacy of a Supervised Home-based Standard Physical Exercise Program, for Metastatic Cancer Patients Receiving Oral Targeted Therapy: The UNICANCER SdS 01 QUALIOR Study
Brief Title: QUALIOR Feasibility and Efficacy of a Supervised Home-based Standard Physical Exercise Program
Acronym: QUALIOR
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: UNICANCER (Other)
Collaborators: CAMI: Sport & Cancer (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: UC-0106/1510 SdS 01 QUALIOR
Record Dates: First submitted 2017-05-22; First posted 2017-05-30 (Actual); Last update posted 2024-11-12 (Actual); Status verified 2024-11

CONDITIONS: Home Based Standardised Adapted Physical Activity Programme; Patients Taking Oral Targeted Therapy for Metastatic Cancer
Keywords: Adapted physical activity; Oral targeted therapy; Advanced cancer; Fatigue; Quality of life; Randomized Study
MeSH Terms: conditions — Fatigue

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ARM A: A (Experimental): Supervised physical exercise programs (SPEP)
  Interventions: Behavioral: Supervised physical exercise programs
- ARM B: B (Active Comparator): Adapted physical activity (APA)
  Interventions: Behavioral: Adapted physical activity

INTERVENTIONS:
Behavioral: Supervised physical exercise programs — A weekly supervised physical activity session of 60 min at the patient's home is planned for 3 months.
  These sessions will be supervised by an educator or physiotherapist trained, with respect to the pathology and the clinical study, specifically for this activity (Fédération Française Sport et Cancer) . The proposed exercises will be normalized and adapted to each patient's profile.
  Self reported questionnaires: FACT-F, FACT-G, EQ-5D, FAACT module AC/S, FACT-Gog, HADS, IPAQ, Evaluation by a coach VAE
  Arms: ARM A: A
Behavioral: Adapted physical activity — Program based on the recommendations for performing a physical activity. A booklet containing physical activity recommendations will be given to the patients after randomization.
  The weekly sessions at the patients home for the experimental group (Program A) must begin as soon as possible within the 15 days after starting oral targeted therapy.
  Self reported questionnaires: FACT-F, FACT-G, EQ-5D, FAACT module AC/S, FACT-Gog, HADS, IPAQ
  Arms: ARM B: B

SUMMARY:
This phase II-III study will be randomized (2:1) patients starting first-line oral targeted therapies (OTT) for metastatic cancer between an individualized supervised physical exercise programs (SPEP) by a personal coach, and recommended physical exercises via a booklet. Eligible patients will have received ≤2 lines of metastatic chemotherapy, Eastern Cooperative Oncology Group Performance status (ECOG PS) ≤2, controlled pain (visual analogue scale (VAS) <3/10), and life expectancy ≥3 months.

ELIGIBILITY:
Inclusion Criteria:

1. Patient's ≥18 years old.
2. Patient treated for a metastatic solid tumour within the following 4 cohorts: breast cancer, kidney cancer, lung cancer, and other tumours treated with oral targeted therapies (including melanomas, sarcomas, hepatic sarcomas, and colon cancers).
3. Patients starting first-line oral targeted therapy, with market authorisation. The targeted therapy may be associated with hormonal therapy.
4. Patients may have been treated with immunotherapy.
5. Patients may have received chemotherapy (≤2 lines) for their metastatic disease.
6. Life expectancy of ≥3 months.
7. ECOG performance status ≤2.
8. Patients able to comply with the constraints of the SPEP protocol.
9. Pain under control (VAS ˂3; 0-10 scale).
10. Haemoglobin level ≥9 g/dL.
11. Patient must have signed the informed consent form before any study-related procedures.
12. Patients must have public health insurance coverage.

Exclusion Criteria:

1. Patient receiving an injectable targeted therapy.
2. Patient previously treated by more than 2 lines of treatment (previous treatment with cytokines are allowed)
3. Patient to be treated with chemotherapy associated with the oral targeted therapy (hormonal therapy is allowed).
4. Patient with known risk of fracture, symptomatic cardiac insufficiency (NYHA-3), respiratory insufficiency (grade 3), intense pain not controlled with analgesic treatment, and/or neuropathy (grade 3).
5. Patients with a history of cancer in the last 5 years (except basal cell carcinoma adequately treated and in situ cervical cancer treated and cured).
6. Patient treated with corticotherapy (˃1 month) before randomisation at a dose ˃1 mg/kg.
7. Bone metastases with risk of fractures.
8. Geographical, sociological, or psychological reasons that could potentially hampering compliance with the study protocol and follow-up schedule.
9. Patients with a history of non-compliance to medical treatment, reluctance or incapable to conform to the study protocol.
10. Persons deprived of liberty or under guardianship.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 190 (Actual)
Dates: Start 2017-07-11 (Actual); Primary Completion 2024-09-30 (Actual); Study Completion 2028-07-11 (Estimated)

PRIMARY OUTCOMES:
FACT-F relative on Fatigue | Month 3 ( M3)
  Self reported Questionnaires
FACT-G | Month3 ( M3)
  Self Reported Questionnaire relative on Well-Being Patient

SECONDARY OUTCOMES:
PFS | From date of randomization until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 75 months
  Progression Free Survival
OS | From date of randomization until the date of first documented date of death from any cause, whichever came first, assessed up to 75 months
  Overall Survival
Quality of life | Month 1, Month 2, Month 3, and every 3 months for 1 year
  Self reported Questionnaire on quality of life
Fatigue | Month 1, Month 2, Month 3, and every 3 months for 1 year
  Self reported Questionnaire FACT-F on Fatigue
Fatigue | Month 1, Month 2, Month 3, and every 3 months for 1 year
  visual analogic scale for fatigue
Pain | Month 1, Month 2, Month 3, and every 3 months for 1 year
  visual analogic scale for pain (VAS)
Toxicities Secondaries effectsToxicities according NCI-CTC (National Cancer Institute Updates CTCAE to v.4.03. Common Terminology Criteria ) | Baseline, Month 1, Month 2, Month 3, and every 3 months for 1 year
  Incidence of Treatment-Emergent Adverse Events [Safety and Tolerability]).
Compliance about oral targeted therapy | Baseline, Month 1, Month 2, Month 3
  Self reported Questionnaire Morisky-Green
Benefit of physical activity: walk | Baseline, Month 1, Month 2, Month 3 and every 3 months for 1 year
  6 minutes walking test
Benefit of physical activity muscle function | Baseline, Month 1, Month 2, Month 3 and every 3 months for 1 year
  muscle function
Benefit of physical activity muscle strength | Baseline, Month 1, Month 2, Month 3 and every 3 months for 1 year
  muscle strength
Physical Activity IPAQ | Baseline, Month 1, Month 2, Month 3 and every 3 months for 1 year
  self reported Questionnaire IPAQ ( International Physical Activity Questionnaire)
Physical Activity, Body Mass Index | Baseline, Month 1, Month 2, Month 3 and every 3 months for 1 year
  Body Mass Index
Scores of anxiety and depression | Baseline, Month 1, Month 2, Month 3
  Hospital Anxiety and Depression Scale (HADs)
Cognitive functions | Baseline, Month 1, Month 2, Month 3 and every 3 months for 1 year
  Self reported questionnaire FACT-Cog
Evaluation of Ingesta, Anorexia | Baseline, Month 3
  Ingesta
Evaluation of Ingesta, VAS | Baseline, Month 3
  VAS
Evaluation of Anorexia | Baseline, Month 1, Month 2, Month 3 and every 3 months for 1 year
  Self reported FAACT (module A-C)

CONTACTS AND LOCATIONS:
Overall Officials: Florence JOLY, MD PhD, Principal Investigator — Centre François Baclesse
Locations (15):
- France (15):
  - ICO Paul Papin, Angers
  - CH Annecy Genevois - site d'Annecy, Annecy
  - CHRU de Besançon, Besançon
  - Centre François Baclesse, Caen
  - CH de Cholet, Cholet
  - GHMG - Institut Daniel Hollard, Grenoble
  - CHD Vendée, La Roche-sur-Yon
  - Hospices Civils de Lyon - Hôpital Louis Pradel, Lyon
  - CHU La Timone, Marseille
  - ICO RenéGauducheau, Nantes
  - CH Nimes - Institut de Cancérologie du Gard, Nîmes
  - Institut Curie Paris, Paris
  - Centre Eugène Marquis, Rennes
  - INSTITUT CURIE - Site René Huguenin St Cloud, Saint-Cloud
  - HIA Begin, Saint-Mandé

IPD SHARING:
Plan to Share IPD: No
Individual Participant Data will not be shared at an individual level. Those data will be part of the study database including all enrolled patients.

REFERENCES:
- [Derived] Joly F, Lefeuvre-Plesse C, Garnier-Tixidre C, Helissey C, Menneveau N, Zannetti A, Salas S, Houede N, Abadie-Lacourtoisie S, Stefani L, Nenan S, Rieger I, Durand-Zaleski I, Descotes JM, Anota A. Feasibility and efficacy of a supervised home-based physical exercise program for metastatic cancer patients receiving oral targeted therapy: study protocol for the phase II/III - UNICANCER SdS 01 QUALIOR trial. BMC Cancer. 2020 Oct 9;20(1):975. doi: 10.1186/s12885-020-07381-4. PMID 33036567